CLINICAL TRIAL: NCT00105313
Title: A Phase I Open-Label Dose Escalation Study to Evaluate MEDI-507 in Patients With CD2-Positive Lymphoma/Leukemia
Brief Title: Study to Evaluate MEDI-507 in Patients With CD2-Positive Lymphoma/Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: After review of safety events and have decided that further dose escalation of MEDI-507 as a single agent is not feasible.
Sponsor: MedImmune LLC (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP107
Record Dates: First submitted 2005-03-11; First posted 2005-03-14 (Estimated); Last update posted 2007-06-14 (Estimated); Status verified 2007-06

CONDITIONS: Lymphoma; Leukemia; Cancer
MeSH Terms: conditions — Lymphoma; Leukemia; Neoplasms | interventions — siplizumab

INTERVENTIONS:
Drug: MEDI-507

SUMMARY:
For primary objectives, we will determine the MTD and examine clinical responses and immune cell populations to determine an OBD, and describe the safety and tolerability of MEDI-507.

For the secondary objectives we will look at the antitumor activity of MEDI 507, PK, serum concentrations, and immunogenicity of MEDI-507, as well as time courses of depletion and recovery of CD2 positive and total T-Cell populations.

ELIGIBILITY:
Individuals may be eligible for this study if they are 18 years of age or older and:

* Have one of the following types of T-Cell Lymphoproliferative disorders such as Cutaneous T-cell Lymphoma (CTCL), Peripheral T-cell Lymphoma (PCTL), Large Cell Lymphoma (LGL), or Adult T-cell Lymphoma (ATL). Patients should have disease that is resistant or refractory to the front-line therapy, except ATL patients for whom there is no standard therapy.
* At least 30% of tumor cells must be CD2 positive.
* Karnofsky Performance status of greater than or equal to 70% (able to care for themselves; but unable to carry on normal activity or to do active work).
* At least 3 weeks must have passed since prior systemic cytotoxic chemotherapy, prolonged or cytolytic steroid therapy or major surgery, and all treatment-related toxicities must have resolved prior to the first MEDI-507 administration (except thrombocytopenia).
* Have no prior treatment with MEDI-507.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-02

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) or the optimal biological dose
(OBD) of MEDI-507 based on safety and tolerability of MEDI-507 in patients with
CD-2 positive lymphoproliferative disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Luz Hammershaimb, MD, Study Director — MedImmune LLC
Locations (11):
- United States (11):
  - USC/Norris Cancer Center, Los Angeles, California
  - Yale Cancer Center, New Haven, Connecticut
  - Georgetown University Medical Center, Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Ctr & Research Institute Div of Hem/Onc, Tampa, Florida
  - University of Maryland School of Medicine, Greenebaum Cancer Center, Baltimore, Maryland
  - Tufts New England Medical Center, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Kimmel Cancer Center, Thomas Jefferson University, Philadelphia, Pennsylvania
  - M.D. Anderson Cancer Center, Houston, Texas